CLINICAL TRIAL: NCT06896643
Title: Urinary Infection and Colonization in Bone Procedures
Status: Recruiting | Type: Observational
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Klára Nekvindová, Deputy Chief for Science, Education, and Research, Tomas Bata Hospital, Czech Republic
Other Study IDs: 2024-32
Record Dates: First submitted 2025-03-04; First posted 2025-03-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Urinary Tract Infection; Complications; Urinary Tract Infection (Diagnosis); Frailty
Keywords: urinary; tract; infection; colonization; postoperative complications
MeSH Terms: conditions — Urinary Tract Infections; Disease; Frailty; Infections; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For seniors aged 65 and over (inclusive) undergoing surgical procedures (bone surgery, traumatology, orthopedics) in an acute or elective setting, the relationship between preoperative urinary tract infection/colonization (within 30 days before the procedure) and the occurrence of predefined postoperative complications (monitoring during the patients' hospitalization) will be observed

DETAILED DESCRIPTION:
For seniors aged 65 and over (inclusive) undergoing surgical procedures (bone surgery, traumatology, orthopedics) in an acute or elective setting, the relationship between preoperative urinary tract infection/colonization (within 30 days before the procedure) and the occurrence of predefined postoperative complications (monitoring during the patients' hospitalization) will be observed Among the monitored parameters before the surgical procedure will be urine collection (chemical + sediment - a common part of the pre-anesthetic examination), and in case of findings, a sample for bacteriological examination will be indicated. Additionally, subjective symptoms (present, absent), presence of fever, whether the infection/finding in the urine was treated or not, and whether a control urine examination was performed (performed, not performed) will be recorded. The origin of the patient (home, social care facility) and the planned surgical procedure will be noted. The Clinical Frailty Scale, type of anesthesia (general, regional), and any administered antibiotic treatment will also be recorded.

After the surgical procedure, the occurrence of urinary infection (yes, no, sample not taken) will be assessed. Postoperative complications such as fever, circulatory instability, development of delirium, infection, septic state, and death will be monitored. The trajectory of the respondent during hospitalization (which departments they will be treated in, including the length of hospitalization) will be recorded. The primary goal will be to determine the relationship between the preoperative occurrence of urinary infection or colonization in patients within the last 30 days before the procedure and the occurrence of predefined postoperative complications. Secondary goals will include identifying the most common postoperative complications in patients with preoperative urinary colonization or proven urinary infection. Additionally, the relationship between the preoperative Clinical Frailty Scale in the defined patient population and the occurrence of predefined postoperative complications will be examined. The final secondary goal will be to determine preoperative antibiotic therapy in the preoperative period.

The cohort of traumatology patients undergoing surgical procedures was chosen to ensure the homogeneity of the studied population (seniors over 65 undergoing bone surgery).

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years, including
* Elective or acute trauma/orthopedic bone surgery
* Urine examination as part of pre-anesthetic examination, urine + sediment, in case of suspicion - bacteriological examination
* Signed informed consent for research as part of pre-anesthetic examination (I or II), respecting informed consent as an expression of the patient's "free will"

Exclusion Criteria:

* Negative finding in urine: chemical examination + sediment preoperatively
* Respondent under the influence of premedication, alcohol, or drugs
* Sensory impairment (blindness)
* Delirious preoperative state
* Severe mental disorder
* Sopor
* coma
* Septic state
* Acute respiratory failure
* Disagreement with participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: For seniors over 65 years (including), undergoing surgery (bone procedure, traumatology, orthopedics) in an acute or elective mode, the relationship between preoperative infection/colonization of the urinary tract (within 30 days before the procedure) and the occurrence of predefined postoperative complications will be monitored.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infection preoperatively - signs and symptoms | one week before surgery
  Signs and symptoms include dysuria, frequency, urgency, or/and fever or/and smelling urine and non-specific signs (nausea, malaise)
Urinary tract infection preoperatively - urinary dipstick test. | one week before surgery
  Positive urine dipstict test (i.e. nitrate-reductace and leukocyte esterase detection).
Urinary tract infection preoperatively - chemical examination of the urine and sediment - pH | one week before surgery
  Positive result in chemical examination of the urine and the sediment for the possibility of infection s: pH ≥ 6.
Urinary tract infection preoperatively: chemical examination - proteinuria (urine dipstick test) | one week before surgery
  Detection of proteinuria with urine dipstick test.
Urinary tract infection preoperatively - leukocytouria (urine dipstick test) | one week before surgery
  Positive result t is leukocyturia (detection of leucocyte esteras) in a dipstick test.
Urinary tract infection preoperatively chemical examination of the urine and sediment -pyuria (urine dipstick test) | one week before surgery
  Pyuria, which is the presence of white blood cells in the urine, will detected through these methods: Postive urine dipstick test - showing leukocyte esterase or nitrites.
  And additionally have to present: discoloration, clouding or change in the smell of urine for a pyuria
Urinary tract infection preoperatively: chemical examination of the urine and sediment -bacteriuria (urine dipstick test) | one week before surgery
  Presence of bacteriuria (presence of bacteria in the urine). Can be detected through urine dipstick test (determination of presence of leukocyte esterase and nitrites, which are indicators of white blood cells and bacteria in the urine)
Urinary tract infection preoperatively - chemical examination preoperatively - chemical examination of the urine and sediment -bacteriuria | one week before surgery
  Presence of bacteriuria (presence of bacteria in the urine). Can be detected through through flow cytometry (this method detects bacteria in urinary samples in the range from 40 up to 1000/μl),
Urinary tract infection preoperatively: chemical examination of the urine and sediment -bacteriuria (urine culture) | one week before surgery
  Presence of bacteriuria (presence of bacteria in the urine). Can be detected through urine culture (bacteria grow from a urine sample, cutoff is for a significant bacterial count is typically greater than 100,000 colony-forming units (CFU) per mililiter).
Urinary tract infection preoperatively - chemical examination preoperatively - chemical examination of the urine and sediment - proteinuria | one week before surgery
  Detection of proteinuria with the sulfosalicylic acid test in laboratory.
  A semiquantitative scale is used for evaluation:
  1. Opalescence - approximate concentration of protein in g/l: 0,05-0,1
  2. Slight turbidity (transparent, underlying text can be read - approximate concentration of protein in g/l: 0,1-0,2
  3. Milky turbidity (opaque, without flakes) - approximate concentration of protein in g/l: 0,5-1,0
  4. Milky turbidity with flake formation: approximate concentration of protein in g/l: 2,0-5,0
  5. Flocculent precipitate: approximate concentration of protein in g/l ≥ 5,0
Urinary tract infection preoperatively - leukocytouria (sediment) | one week before surgery
  Positive result is finding in the in sediment more than 10 leukocytes per field of view.
Urinary tract infection preoperatively chemical examination of the urine and sediment -pyuria (microscopy) | one week before surgery
  Pyuria, which is the presence of white blood cells in the urine, will detected through these methods: Microscopy - cell counts performer by microscopy, positive finding is more than 10 leukocytes per field of view.
  And additionally have to present: discoloration, clouding or change in the smell of urine for a pyuria.
Urinary tract colonization preoperatively - asymptomatic bacteriuria, women (urine culture) | one week before surgery
  Midstream clean catch urine specimen will be needed. Two consecutive specimens with isolation of the same bacteria species with at least 100,000 colony-forming units (CFUs) per ml of urine.
Urinary tract colonization preoperatively - asymptomatic bacteriuria, men (urine culture) | one week before surgery
  Midstream clean catch urine specimen will be needed. For men, a single specimen with isolation of one bacteria species with at least 100,000 CFUs per ml of urine.
Urinary tract colonization preoperatively - asymptomatic bacteriuria, catheterized specimen (urine culture)) | one week before surgery
  For women or men, a single specimen with isolation of one bacteria species with at least 100 CFUs per ml of urine.
Antibiotic therapy before the surgery | one week before surgery
  Preoperative antibiotic use will be recorded. Options yes, no. If yes, the type of antibiotic used will be recorded.
Postoperative complications - fever | one week after surgery
  Fever is defined as a body temperature above 38 degrees Celsius
Postoperative complications -circulatory instability | one week after surgery
  Presence of hypotension, MAP below 70 mm Hg
Postoperative complications -I nfection | one week after surgery
  Presence of infection and origin of the infection in laboratory findings and in clinical picture.
Postoperative complications - sepsis | one week after surgery
  Presence of sepsis and origin of the infection in laboratory findings and in clinical picture.
Postoperative complications -postoperative delirum | one week after surgery
  Presence of postoperative delirium. To determine the diagnose CAM-ICU will be used.
Postoperative complications - antibiotic | one week after surgery
  Administered antibiotic treatment and its duration

SECONDARY OUTCOMES:
Clinical frailty scale (CFS) preoperatively | one week before surgery
  The CFS is a nine-point scale based on clinical evaluation of mobility, energy, physical activity, and function.
  Clinical Frailty Scale Components: 1. Very fit, 2. Well, 3. Managing Well:, 4. Living With Very Mild Frailty, 5. Living with Mild Frailty: 6. Living With Moderate Frailty, 6. Living With Severe Frailty, 8. Living with Very Severe Frailty, 9. Terminally Ill
Preoperative antibiotic therapy | one week before surgery
  Preoperatively, it will be assessed whether the patient received antibiotic treatment for a urinary tract infection prior to surgery. The result will be recorded as yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Tomas Bata Hospital, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parvizi J, Koo KH. Should a Urinary Tract Infection Be Treated before a Total Joint Arthroplasty? Hip Pelvis. 2019 Mar;31(1):1-3. doi: 10.5371/hp.2019.31.1.1. Epub 2019 Mar 5. PMID 30899708

DOCUMENTS (1):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT06896643/Prot_000.pdf